CLINICAL TRIAL: NCT06743763
Title: Comparative Effectiveness of fNIRS-Based Neurofeedback Training in Children With ADHD: The Impact of Virtual Reality Integration
Brief Title: fNIRS-Based Neurofeedback Training in Children With ADHD: The Effects of VR
Acronym: VR-fNIRS-RCT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kathy Shum, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA200247(RCT2)
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: neurofeedback; fNIRS; ADHD; children; virtual reality
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Experimental group: receives 8-week functional near-infrared spectroscopy (fNIRS) neurofeedback training (coupled with virtual reality), twice per week, each lasting 1 hour.
  Comparative group 1: receives 8-week functional near-infrared spectroscopy (fNIRS) neurofeedback training without virtual reality(VR) technology, twice per week, each lasting 1 hour.
  Comparative group 2: receives 8-week training using VR technology (without neurofeedback) twice per week, each lasting 1 hour.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fNIRS-NFT with VR (Experimental): The experimental group will receive 16 sessions of training, 1 hour each, conducted twice per week over a period of 8 weeks. A classroom setting will be stimulated using VR and participants will be asked to complete some academic-related tasks during the stimulated lessons. The sensor on the neurofeedback device worn by the participants will detect changes in the blood oxy-hemoglobin level in brain cortical tissue and feedback to the participants via visual images or auditory sounds from the computer. Through practice, participants will learn to manipulate their attention, presumably by altering brain activities.
  Interventions: Behavioral: fNIRS-based neurofeedback; Behavioral: Virtual Reality Simulated Classroom
- fNIRS-NFT without VR (Active Comparator): The fNIRS-NFT without VR (NFT-2D group) will receive 16 sessions of training, 1 hour each, conducted twice per week over a period of 8 weeks. A classroom setting will be stimulated via a computer screen and participants will be asked to complete some academic-related tasks during the stimulated lessons by pressing a remote controller provided. The sensor on the neurofeedback device worn by the participants will detect changes in the blood oxy-hemoglobin level in brain cortical tissue and feedback to the participants via visual images or auditory sounds from the computer. Through practice, participants hopefully will learn to manipulate their attention, presumably by altering brain activities.
  Interventions: Behavioral: fNIRS-based neurofeedback
- VR without fNIRS-NFT (Active Comparator): In the VR without fNIRS-NFT Training, we have designed a virtual reality classroom scenario modeled and children are asked to complete academic tasks in the VR setting but no neurofeedback will be provided.
  Interventions: Behavioral: Virtual Reality Simulated Classroom

INTERVENTIONS:
Behavioral: fNIRS-based neurofeedback — fNIRS-based neurofeedback is provided during a simulated classroom scenario where the child participants are asked to learn to regulate their attention based on the feedback provided by the fNIRS on the oxygenated haemoglobin level in their prefrontal cortex.
  Arms: fNIRS-NFT with VR; fNIRS-NFT without VR
Behavioral: Virtual Reality Simulated Classroom — A simulated classroom scenario is integrated in VR setting and children are asked to complete academic tasks in the simulated classroom.
  Arms: VR without fNIRS-NFT; fNIRS-NFT with VR

SUMMARY:
The study aims to explore whether the treatment using fNIRS-based neurofeedback training for children with attention-deficit/hyperactivity disorder (ADHD) is useful. Furthermore, the study hopes to evaluate whether the use of virtual reality (VR) technology will have an impact on the treatment's effectiveness.

The program includes the following components:

Participants will be randomly assigned to one of three intervention groups: the neurofeedback with virtual reality (VR) group, the 2D neurofeedback group (with no VR technology applied), and the VR without neurofeedback group. All participants will complete academic-related tasks in simulated lessons. Participants in the VR neurofeedback group will wear VR goggles and a neurofeedback device that measures blood oxy-hemoglobin levels in brain cortical tissue and provides feedback via visual images or auditory sounds to the participants. Those in the 2D neurofeedback group will use a computer to complete the tasks, with all other settings (e.g., neurofeedback settings) remaining the same. The VR without neurofeedback group will wear VR goggles to complete tasks, but without the neurofeedback component.

All participants will complete a total of 16 training sessions over 8 weeks (twice a week), with each session lasting approximately 35 to 60 minutes.

To investigate the intervention's effectiveness, children will be asked to complete a set of cognitive tests covering inhibitory control, attention, and working memory before the intervention (i.e., Time 1), immediately after the 8-week training (i.e., Time 2), and 2 months after the training (i.e., Time 3, a 2-month follow-up). The assessment will take around 1 hour and will be conducted at the laboratory at the University of Hong Kong. Additionally, parents and teachers will be asked to complete a questionnaire assessing children's behavior at home and at school at three time points.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7- 12
* Clinical diagnosis of ADHD
* Significant teacher- or parent-reported attention problems during screening

Exclusion Criteria:

* Inability to answer the first five questions in Raven's Progressive Matrices
* Hearing, visual, or physical impairments that might hinder participation in the training and assessment activities
* Clinical diagnosis and suspected cases of Autism Spectrum Disorder (ASD)
* Prior or current participation in NFT
* Current participation in a psychotherapeutic treatment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Children's ADHD symptoms | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  Parents will be asked to complete the Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) measuring children's inattentive, hyperactive and impulsive symptoms with a 4-point Likert scale (ranges from 0 to 3). The minimum total score is 0 while the maximum total score is 78, with a higher score indicating a higher level of inattentive, hyperactive and impulsive symptoms.
Children's ADHD symptoms | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Parents will be asked to complete the Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) measuring children's inattentive, hyperactive and impulsive symptoms with a 4-point Likert scale (ranges from 0 to 3). The minimum total score is 0 while the maximum total score is 78, with a higher score indicating a higher level of inattentive, hyperactive and impulsive symptoms.
Children's ADHD symptoms | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  Parents will be asked to complete the Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) measuring children's inattentive, hyperactive and impulsive symptoms with a 4-point Likert scale (ranges from 0 to 3). The minimum total score is 0 while the maximum total score is 78, with a higher score indicating a higher level of inattentive, hyperactive and impulsive symptoms.

SECONDARY OUTCOMES:
Conners Continuous Performance Test 3rd Edition (CPT 3) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Conners Continuous Performance Test 3rd Edition (CPT 3) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Conners Continuous Performance Test 3rd Edition (CPT 3) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Functional NIRS | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured during the direct assessment task of Conners Continuous Performance Test 3rd Edition (CPT3) using functional NIRS.
Functional NIRS | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured during the direct assessment task of Conners Continuous Performance Test 3rd Edition (CPT3) using functional NIRS.
Functional NIRS | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured during the direct assessment task of Conners Continuous Performance Test 3rd Edition (CPT3) using functional NIRS.
Number subtest of Children's Memory Scale (CMS) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Number subtest of Children's Memory Scale (CMS) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Number subtest of Children's Memory Scale (CMS) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Behavioural ratings on children's executive functions | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  Parents and teachers will be asked to complete Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation
Behavioural ratings on children's executive functions | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Parents and teachers will be asked to complete Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation
Behavioural ratings on children's executive functions | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  Parents and teachers will be asked to complete Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation

OTHER OUTCOMES:
Children's enjoyment of the training | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Children's enjoyment of the training will be evaluated using the Cognitive Absorption Scale (CAS) using a 7-point Likert scale (ranges from 1 to 7), which includes four dimensions: temporal dissociation, focused immersion, heightened enjoyment, and curiosity. The total score of this scale ranges from 7 to 119, with a higher score indicating a higher level of children's enjoyment of the training.
Feasibility of conducting VR training within children | Up to 8 to 10 weeks (within the intervention period)
  Children's symptoms of cybersickness (e.g., nausea, fatigue, eye strain) will be measured using the Simulator Sickness Questionnaire (SSQ) after completing every training session, using a 4-point Likert scale (ranges from 0 to 3). The minimum weighted total score of this scale is 0 and the maximum weighted total score is 235.62, with a higher score indicating a higher level of symptoms of cybersickness.

CONTACTS AND LOCATIONS:
Overall Officials: Kar-man Kathy Shum, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be available upon reasonable request.
Time Frame: Beginning immediately after publication and ending 5 years after publication.
Access Criteria: To gain access, requestors will need to provide a clear research aim or methodological sound research plan directed to the principal investigator (kkmshum@hku.hk).